CLINICAL TRIAL: NCT01558739
Title: A UK Open-label, Multicentre, Exploratory Phase II Study of INC424 for Patients With Primary Myelofibrosis (PMF) or Post Polycythaemia Myelofibrosis (PPV MF) or Post Essential Thrombocythaemia Myelofibrosis (PET-MF)
Brief Title: Exploratory Phase II Study of INC424 Patients With Primary Myelofibrosis (PMF) or Post Polycythaemia Myelofibrosis (PPV MF) or Post Essential Thrombocythaemia Myelofibrosis (PET-MF)
Acronym: MACS2030
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424AGB02; 2011-005066-38 (EudraCT Number)
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Results first posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Primary Myelofibrosis (PMF); Post Polycythaemia Myelofibrosis (PPV MF); Post Essential Thrombocythaemia Myelofibrosis (PET-MF)
Keywords: Ruxolitinib; INC424; myelofibrosis; PMF; post polycythemia myelofibrosis; PPV MF; post-essential thrombocythemia myelofibrosis; PET-MF; Primary Myelofibrosis; Polycythemia; Thrombocythemia; Essential Thrombocytosis; myeloproliferative Disorders; Bone Marrow Diseases; Haematologic Diseases; Blood Coagulation Disorders; Blood Platelet Disorders; Haemorrhagic Disorders
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia; Thrombocytosis; Thrombocythemia, Essential; Myeloproliferative Disorders; Bone Marrow Diseases; Blood Coagulation Disorders; Blood Platelet Disorders; Hemorrhagic Disorders | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INC424 (Experimental): Patients diagnosed with PMF, PPV MF, or PET-MF were treated with oral INC424 at a dose of 15 - 20 mg (dose based on Baseline platelet count) twice daily.
  Interventions: Drug: INC424

INTERVENTIONS:
Drug: INC424 — Ruxolitinib was provided in 5 mg tablets, packaged in bottles. 15 - 20 mg (dose based on Baseline platelet count) twice daily.

SUMMARY:
The primary objective of this study is to evaluate the efficacy of INC424 in patients with PMF, PPV MF, or PET-MF using a composite measure of either an objective endpoint (> 50% reduction in splenomegaly using palpitation at 48 weeks) and/or a subjective endpoint (>50% reduction in total symptom score at 48 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients must not be eligible for another ongoing INC424 clinical trial.
* Patients must be diagnosed with PMF, PPV MF or PET-MF, according to the 2008 revised World Health Organization criteria irrespective of JAK2 mutation status.
* Patients with PMF requiring therapy must be classified as high risk (3 prognostic factors) OR intermediate risk level 2 (2 prognostic factors, no more), OR intermediate risk level 1 (1 prognostic factor, no more) with an enlarged spleen. The prognostic factors, defined by the International Working Group are:

  1. Age > 65 years;
  2. Presence of constitutional symptoms (weight loss, fever, night sweats); marked anemia (Hgb < 10g/dL)*;
  3. Leukocytosis (history of WBC > 25 x109/L);
  4. Circulating blasts > 1%. • A hemoglobin value < 10 g/dL must be demonstrated during the Screening Visit for patients who are not transfusion dependent. Patients receiving regular transfusions of packed red blood cells will be considered to have hemoglobin < 10 g/dL for the purpose of evaluation of risk factors.
* Patients with Intermediate-1 disease and splenomegaly must have a palpable spleen measuring 5 cm or greater from the costal margin to the point of greatest splenic protrusion.
* Patients must have a peripheral blood blast count of < 10%.
* Patients with adequate liver function defined as direct bilirubin ≤ 2.0 x ULN and ALT ≤ 2.5 x ULN.
* Patients with adequate renal function defined as serum creatinine ≤ 2 x ULN.
* Patients with an ECOG performance status of 0, 1, or 2 (Appendix 5).

Exclusion criteria:

* Patients eligible for hematopoietic stem cell transplantation (suitable candidate and a suitable donor is available).
* Patients with history of malignancy in past 3 years except for treated, early-stage squamous or basal cell carcinoma in situ.
* Patients undergoing treatment with hematopoietic growth factor receptor agonists (i.e., erythropoietin [Epo], granulocyte colony stimulating factor (GCSF [Neupogen; Neulasta], romiplostim, eltrombopag) at any time within 2 weeks prior to Screening or 4 weeks prior to Baseline.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral INC424 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).
* Patients with cardiac disease which in the Investigator's opinion may jeopardize the safety of the patient or the compliance with the protocol.
* Patients with clinically significant bacterial, fungal, parasitic or viral infection which require therapy. Patients with acute bacterial infections requiring antibiotic use should delay screening/enrollment until the course of antibiotic therapy has been completed.
* Patients with known active hepatitis A, B, C or who are HIV-positive.
* Patients with inadequate bone marrow reserve as demonstrated by:

  1. Absolute neutrophil count (ANC) that is ≤ 1000/µL.
  2. Platelet count that is < 100,000/µL without the assistance of growth factors, thrombopoietic factors or platelet transfusions.
* Patients with any history of platelet counts < 50,000/µL or ANC < 500/µL except during treatment for a myeloproliferative disorder or treatment with cytotoxic therapy for any other reason.
* Patients with coagulation parameters (PT, PTT, INR) ≥ 1.5.
* Patients with known hypersensitivity to INC424 or other JAK1/2 inhibitors, or to their excipients.
* Patients under ongoing treatment with another investigational medication or having been treated with an investigational medication within 30 days of screening.
* Patients with any concurrent condition that, in the Investigator's opinion would jeopardize the safety of the patient or compliance with the protocol.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Novartis Pharmaceuticals
Locations (9):
- United Kingdom (9):
  - Novartis Investigative Site, Cardiff, Wales
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, East Yorkshire
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Oxford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 54 patients were screened. 48 patients were enrolled as planned.
Period: Overall Study
Arm/Group | INC424
Started | 48
Completed | 31
Not Completed | 17
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 2
Not completed — Death | 3
Not completed — Disease Progression | 4
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients were included in the Full Analysis Set and the Safety Set.
Arm/Group | INC424
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.12 (10.419)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Success
Description: Treatment success was defined as a 50% or greater reduction in palpable spleen length versus baseline at 48 weeks and/or a 50% or greater improvement in total symptom score (derived from the MF symptom assessment form (MFSAF) questionnaire) versus baseline at the week 48 time point. The MFSAF assesses the following symptoms (all scored from absent (0) to worst imaginable (10)): general fatigue, abdominal pain (and discomfort), inactivity (ability to move and walk around), cough, night sweats, itching (pruritus), bone pain (diffuse not joint pain or arthritis), fever, change in appetite/unintentional weight loss (or gain) in past 6 months, overall quality of life (QoL).
Time Frame: 48 Weeks
Population: Full analysis set (FAS): The FAS included all participants who received at least one administration of study drug and had at least one post-baseline efficacy assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | INC424
Number analyzed (Participants) | 48
Percentage of participants | 50

2. Secondary Outcome: Percentage of Participants With Best Overall Response
Description: Response to treatment and disease progression was assessed by physical examination, specifically assessing changes in spleen size by palpation. Disease response and progression was evaluated using the International Working Group for myelofibrosis Research and Treatment Response Criteria.
Time Frame: week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | INC424
Number analyzed (Participants) | 48
Percentage of participants
  Clinical improvement | 6.3
  Complete response | 6.3
  Partial response | 39.6
  Stable disease | 47.9

3. Secondary Outcome: Change From Baseline in Myelofibrosis Symptoms Assessment Form (MF-SAF)
Description: The MF-SAF consists of seven questions about key symptoms and impact of MF. Questions are scored on a scale of 0-10, with higher scores indicating more severe symptoms and greater inactivity. Questions 1-6, which together comprise a Total Symptom Score (TSS), investigate the following symptoms: night sweats, pruritus/itching, abdominal discomfort, pain under the ribs, early satiety and bone/muscle pain. Question 7 asks patients to report levels of inactivity. The TSS reflects the sum of the scores of these symptoms excluding inactivity, with the maximum possible score being 60 (most severe symptom experienced).
Time Frame: Baseline, week 4, week 12, week 24, week 48
Population: Only participants from the full analysis set (FAS), who had evaluable measurements at both baseline and the post-baseline week time point, was included in the analysis for that time point. The FAS included all participants who received at least one administration of study drug and had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | INC424
Number analyzed (Participants) | 48
score on a scale
  Week 4 (n=37) | -8.78 (10.638)
  Week 12 (n=35) | -8.46 (12.871)
  Week 24 (n=30) | -9.13 (11.950)
  Week 48 (n=18) | -7.83 (9.966)

4. Secondary Outcome: Change From Baseline in EQ5D Preference Index (5 Level EuroQol Questionnaire Determining Quality of Life) From Baseline
Description: The EQ-5D is a standardized instrument used for measuring health outcomes in a wide range of health conditions and treatment. It consists of a descriptive system and a visual analogue scale (EQ-VAS). The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The EQ-VAS records the participant's self-rated health on a vertical, VAS where the endpoints are labeled 'best imaginable health state' and 'worst imaginable health state'. The EQ-5D health state was converted to a single summary index by applying a formula that attaches a weight to each of the levels in each dimension. The final EQ5D preference index scores range from 0 to 1 with higher scores indicating better health.
Time Frame: Baseline, week 4, week 12, week 24, week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | INC424
Number analyzed (Participants) | 48
unit on a scale
  week 4 (n=40) | 0.06 (0.173)
  week 12 (n=38) | 0.05 (0.178)
  week 24 (n=34) | 0.05 (0.231)
  week 48 (n=29) | 0.03 (0.222)

5. Secondary Outcome: Number of Hospitalizations
Description: Medical resource utilization (MRU) was assessed according to the number of hospitalizations.
Time Frame: week 12, week 24, week 26, week 48
Population: Only participants from the full analysis set (FAS), who had evaluable measurements at the post-baseline week time point, were included in the analysis for that time point. The FAS included all participants who received at least one administration of study drug and had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: number of hospitalizations
Arm/Group | INC424
Number analyzed (Participants) | 48
number of hospitalizations
  week 12 (n=48) | 0.10 (0.371)
  week 24 (n=40) | 0.03 (0.158)
  week 36 (n=37) | 0.05 (0.229)
  week 48 (n=35) | 0.09 (0.284)

6. Secondary Outcome: Duration of Hospitalizations
Description: MRU was assessed according to the mean duration of hospitalization visits.
Time Frame: week 48
Population: Participants from the full analysis set, who were hospitalized between baseline and week 48, were included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | INC424
Number analyzed (Participants) | 9
days | 9.00 (5.852)

7. Secondary Outcome: Number of Accident & Emergency Visits From Baseline
Description: MRU was assessed according to the number of accidents and emergency room visits.
Time Frame: baseline to week 12, week 12 to week 24, week 24 to week 36, week 36 to week 48
Population: Only participants from the full analysis set (FAS), who had evaluable measurements at each timeframe, e.g. from baseline to week 12, were included in the analysis for that timeframe. The FAS included all participants who received at least one administration of study drug and had at least one post-baseline efficacy assessment.
Measure: Median (Full Range); unit: Number of visits
Arm/Group | INC424
Number analyzed (Participants) | 48
Number of visits
  baseline to week 12 (n=48) | 0.00 (0.412) [0.0 to 2.0]
  week 12 to week 24 (n=39) | 0.00 (0.160) [0.0 to 1.0]
  week 24 to week 36 (n=33) | 0.00 (0.415) [0.0 to 2.0]
  week 36 to week 48 (n=33) | 0.00 (0.242) [0.0 to 1.0]

8. Secondary Outcome: Number of General Practitioner (GP), Specialists' and Urgent Care Visits
Description: MRU was assessed according to the number of GP, specialists', and urgent care visits.
Time Frame: baseline to week 12, week 12 to, week 24, week 24 to week 36, week 36 to week 48
Population: as for outcome 7
Measure: Median (Full Range); unit: number of visits
Arm/Group | INC424
Number analyzed (Participants) | 48
number of visits
  GP visits, baseline to week 12 (n=45) | 0.0 [0.0 to 4.0]
  GP visits, week 12 to week 24 (n=36) | 0.0 [0.0 to 1.0]
  GP visits, week 24 to week 36 (n=33) | 0.0 [0.0 to 2.0]
  GP visits, week 36 to week 48 (n=33) | 0.0 [0.0 to 3.0]
  Specialists visits, baseline to week 12 (n=47) | 0.00 [0.0 to 8.0]
  Specialists visits, week 12 to week 24 (n=36) | 0.00 [0.0 to 2.0]
  Specialists visits, week 24 to week 36 (n=33) | 0.00 [0.0 to 4.0]
  Specialists visits, week 36 to week 48 (n=33) | 0.00 [0.0 to 3.0]
  Urgent care visits, baseline to week 12 (n=48) | 0.00 [0.0 to 1.0]
  Urgent care visits, week 12 to week 24 (n=39) | 0.00 [0.0 to 0.0]
  Urgent care visits, week 24 to week 36 (n=33) | 0.00 [0.0 to 1.0]
  Urgent care visits, week 36 to week 48 (n=33) | 0.00 [0.0 to 1.0]

9. Secondary Outcome: Percentage of Participants With Transfusion Dependency Status
Description: Transfusion dependency status from baseline through the end of study was assessed. New onset of transfusion dependency was defined as the use of 2 or more units of red blood cell products during the 8 weeks prior to a study visit. New onset of transfusion independency was defined as the use of 0 or 1 unit of red blood cell products during the 8 weeks prior to a study visit.
Time Frame: baseline (BL), end of treatment (up to 28 days post last treatment) (EOT)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | INC424
Number analyzed (Participants) | 48
Percentage of participants
  From independency at BL to independency at EOT | 0.0
  From dependency at BL to independency at EOT | 2.1
  From missing at BL to independency at EOT | 0.0
  From independency at BL to dependency at EOT | 0.0
  From dependency at BL to dependency at EOT | 10.4
  From missing at BL to dependency at EOT | 35.4
  From independency at BL to missing at EOT | 0.0
  From dependency at BL to missing at EOT | 0.0
  From missing at BL to missing at EOT | 52.1

ADVERSE EVENTS:
Arm/Group | INC424
Serious Adverse Events (participants affected / at risk) | 23/48
Other Adverse Events (participants affected / at risk) | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INC424 (N=48)
Anaemia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hernia (General disorders) | 1
Pyrexia (General disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 1
Kidney infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Disorientation (Psychiatric disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Cataract operation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | INC424 (N=48)
Anaemia (Blood and lymphatic system disorders) | 20
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 11
Mouth ulceration (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 11
Pyrexia (General disorders) | 5
Lower respiratory tract infection (Infections and infestations) | 7
Nasopharyngitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 8
Contusion (Injury, poisoning and procedural complications) | 11
Fall (Injury, poisoning and procedural complications) | 6
Alanine aminotransferase increased (Investigations) | 4
Platelet count decreased (Investigations) | 3
Weight increased (Investigations) | 3
Gout (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 9
Headache (Nervous system disorders) | 11
Lethargy (Nervous system disorders) | 10
Paraesthesia (Nervous system disorders) | 3
Depression (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12
Alopecia (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Night sweats (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.